CLINICAL TRIAL: NCT05557227
Title: Galactose - the Ideal Carbohydrate Supplement for Exercise in Type 1 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Principal Investigator, Rakel Johansen, Principal investigator, MD, Ph.D., University of Aarhus
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 93696
Record Dates: First submitted 2022-08-15; First posted 2022-09-27 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Type1diabetes; Hypoglycemia; Hyperglycemia
MeSH Terms: conditions — Hypoglycemia; Hyperglycemia

STUDY DESIGN:
Intervention Model Description: The study is a single-blinded, randomized crossover study, consisting of 4 study days of 1-hour fixed intensity cycling, after consumption of either galactose, lactose, glucose or water.
Who Masked: Participant
Masking Description: The participants will receive either dextrose, water, lactose, galactose in a randomized order (computer generated block randomization) prior to a one-hour exercise bout. Participants, but not investigators, are masked to nutrition allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Galactose (Experimental): 30 g in 200 ml liquid
  Interventions: Other: 1-hour cycling
- Lactose (Experimental): 30 g in 200 ml liquid
  Interventions: Other: 1-hour cycling
- Dextrose (Experimental): 30 g in 200 ml liquid
  Interventions: Other: 1-hour cycling
- Water (Experimental): 200 ml liquid sweetened
  Interventions: Other: 1-hour cycling

INTERVENTIONS:
Other: 1-hour cycling — 60 % VO2 max

SUMMARY:
In this study, 14 subjects with type 1 diabetes are studied in a randomized crossover study in which the subjects cycle at a fixed intensity at 60% of their maximum oxygen capacity (VO2 max) for 1 hour. Thirty minutes before each cycling test, participants consume a 200 ml beverage, consisting of either: 1) dextrose (20 g), 2) galactose (20 g), 3) lactose (20 g) or 4) water (sweetened). If blood sugar drops below 3.9 mmol/l, glucose infusion is given and blood sugar is kept just above 5 mmol/L.

The trial days take place at least 4 days apart.

DETAILED DESCRIPTION:
On study days, a catheter is placed in two antecubital veins for regular blood sampling and for glucose infusion (if needed). The participant will rest in a bed, when not performing the 1-hour bicycle ergometer test.

Thirty minutes before the leg-cycle ergometer test, the participants consume a 300 ml beverage containing either: 1) dextrose (20 g), 2) galactose (20 g) 3) lactose (20 g) or 4) water (sweetened). At t=0, the ergometer test is started and continued for 1 hour (fixed intensity cycling at 60% of VO2-max). If blood glucose drops below 3.9 mmol/l, glucose infusion (5 % glucose) will be administered, and blood glucose is kept just above 5 mmol/l and infused volume is registered.

Blood samples are collected at t= -40, 0, 30, 60, 90, 120 for measurement of plasma lactate, non-esterified fatty acids (NEFA), plasma triglyceride and hormonal concentrations (epinephrine, norepinephrine, cortisol, and glucagon). Plasma blood glucose measurements are performed at t = -40 and every 10-15 minutes until the end of the study day.

Respiratory exchange ratio is measured by indirect calorimetry (collection of respiratory gasses VO2 and VCO2) pre-exercise, at the end of the exercise bout, and 30 minutes post-exercise. Protein oxidation rate is estimated from urinary urea excretion, and net lipid and glucose oxidation rates are calculated from indirect calorimetry measurements with correction for protein oxidation. Therefor a urine sample will also be collected at the end of the study day.

The bicycle ergometer test is discontinued after 1 hour of bicycling and the participant is observed until 2 hour post exercise where the study day is ended.

ELIGIBILITY:
Inclusion Criteria:

* type 1 diabetes for at least 2 years
* age between 18 and 65 years
* HbA1c less than 70 mmol/mol
* Physically active (at least 150 minutes of moderate-to-vigorous intensity activity weekly)
* Insulin pen and pump treatment
* Men and women are eligible, but women will have to perform study days in the mid-cycle phase of the menstrual cycle.

Exclusion Criteria:

* - Diabetic nephropathy, neuropathy, and proliferative retinopathy
* Hypoglycemia unawareness
* Lactose intolerance
* Heart disease and other conditions which may be negatively affected by the VO2 max test and 1-hour cycling on study days

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Time to hypoglycemia Secondary endpoints: Blood glucose variability, volume of intravenous glucose needed to maintain glucose above 5 mmol/l, respiratory exchange ratio. | during and 2 hours after the bicycle test
  time to blood glucose < 3.9 mmol/l

SECONDARY OUTCOMES:
Blood glucose variability | during and 2 hours after the bicycle test
  Change in blood glucose (mmol/l) over time
Glucose infusion | during and 2 hours after the bicycle test
  Volume of intravenous glucose needed to maintain glucose above 5 mmol/l
Respiratory exchange ratio | prior, during and 2 hours after the bicycle test
  RER is measured to to assess carbohydrate and lipid metabolism
Time in Range | prior, during and 2 hours after the bicycle test
  Time spend with a blood glucose between 3,9 mmol/l and 10 mmol/l

CONTACTS AND LOCATIONS:
Locations (1):
- Steno Diabetes Center Aarhus, Aarhus, Region Midt, Denmark

IPD SHARING:
Plan to Share IPD: No